CLINICAL TRIAL: NCT00114530
Title: A Randomized, Open-Label, Phase II Multicenter Study of High-Dose Immunosuppressive Therapy Using Total Body Irradiation, Cyclophosphamide, ATGAM, and Autologous Transplantation With Auto-CD34+HPC Versus Intravenous Pulse Cyclophosphamide for the Treatment of Severe Systemic Sclerosis (SCSSc-01)
Brief Title: Scleroderma: Cyclophosphamide or Transplantation
Acronym: SCOT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT SCSSc-01; NIAID CRMS ID#: 20133 (Other: DAIT NIAID); NCT00472277 (obsolete NCT alias); NCT00545038 (obsolete NCT alias); NCT00848614 (obsolete NCT alias); NCT00871221 (obsolete NCT alias); NCT00872508 (obsolete NCT alias)
Record Dates: First submitted 2005-06-15; First posted 2005-06-16 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Scleroderma, Systemic; Sclerosis; Autoimmune Disease
Keywords: systemic sclerosis; hematopoietic stem cell transplant; clinical trial; global rank composite score
MeSH Terms: conditions — Scleroderma, Systemic; Sclerosis; Autoimmune Diseases | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mHSCT (Experimental): Myeloablative Hematopoietic Stem Cell Transplant (mHSCT) Participants will first have hematopoietic stem cells removed from their blood. They then will receive high doses of chemotherapy and radiation to eliminate their developed and presumably abnormal immune system, followed by autologous stem cell transplantation to reintroduce the purified stem cells to re-establish their immune system.
  Interventions: Biological: mHSCT
- cyclophosphamide (Experimental): Cyclophosphamide (CY) Participants will receive high doses of intravenous cyclophosphamide. The dose being used in this study is about 50% higher than that commonly used by most physicians to treat many other autoimmune diseases.
  Administration of 12 monthly pulses of high-dose intravenous cyclophosphamide (an initial dose of 500 mg/m^2, followed by 11 doses of 750 mg/m^2).
  Interventions: Drug: cyclophosphamide

INTERVENTIONS:
Biological: mHSCT — Hematopoietic progenitors were mobilized with G-CSF. After leukapheresis and CD34+ cell enrichment, the autologous product was cryopreserved. Fractionated TBI (800 cGy), CY (120 mg/kg) and equine antithymocyte globulin (90 mg/kg) were administered as previously reported (References provided in citation section of this ClinicalTrials.gov record: PubMed ID: 17452515 citation and 2.) PubMed ID: 12176878 citation).
  Other Names: Myeloablative Hematopoietic Stem Cell Transplant
  Arms: mHSCT
Drug: cyclophosphamide — An initial intravenous dose of 500 mg/m^2 was followed by 11 infusions of 750 mg/m^2 with mesna given for bladder protection.
  Other Names: cytoxan; CY
  Arms: cyclophosphamide

SUMMARY:
SCOT is a clinical research study designed for people with severe forms of scleroderma. SCOT stands for Scleroderma: Cyclophosphamide Or Transplantation. The SCOT study will compare the potential benefits of stem cell transplant and high-dose monthly cyclophosphamide (Cytoxan) in the treatment of scleroderma.

DETAILED DESCRIPTION:
Severe systemic sclerosis (SSc) is a serious autoimmune disorder in which a person's own immune cells attack organs in the body. SSc affects the skin, joints, lungs, heart, intestinal tract, and kidneys, and half of the patients with the most severe organ involvement die within 5 years. Treatment for SSc usually includes supportive care or immunosuppressive drugs (drugs to suppress the immune system). As the immune cells are believed to be causing the disease, researchers are looking for new therapies that either slow down or stop this process, while not being too toxic.

The main purpose of this study is to determine the safety and effectiveness of high-dose immunosuppressive therapy followed by reinfusion (transplantation) of the participant's own autologous (self) peripheral blood stem cells (PBSCs) compared to treatment with monthly (for 12 months) intravenous doses of cyclophosphamide (Cytoxan) therapy for the treatment of severe systemic sclerosis (SSc). These treatments are being given in order to determine if they will slow down or stop SSc from becoming more severe, and if they can reverse the effects of the disease. The researchers are evaluating the effects of the two treatments on serious organ damage and survival related to SSc, while also looking at the side effects of the two treatments.

This trial also includes three optional mechanistic sub-studies open to a subset of participants enrolled in the SCOT trial:

1. Pharmacokinetics of 4-hydroxycyclophosphamide in Patients Receiving Cyclophosphamide for the SCOT trial (Originally listed separately as DAIT SCSSc-01-01, NCT00848614). The purpose of this study is to determine the plasma concentration and exposure time required for cyclophosphamide to produce optimal immunosuppressive activity with minimal toxicity in participants with severe systemic sclerosis.
2. Vascular Progenitor Cells and the Pathogenesis of Systemic Sclerosis(Originally listed separately as DAIT SCSSc-01-02, NCT00871221). The purpose of this study is to measure and characterize the circulating endothelial progenitor cells from the blood of 30 participants and also to determine the extent of vascular cell apoptosis and proliferation in cutaneous microvasculature in these participants before and after the receipt of the two SCOT treatment regimens.
3. Molecular Analysis of T Cell Immune Recovery for the SCOT Trial(Originally listed separately as DAIT SCSSc-01-03, NCT00872508). The purpose of this study is [1] to describe the condition of peripheral T cell reactivity and repertoire diversity in SSc patients and evaluate evidence for potential defects prior to randomization, [2] to gain a better understanding of the impact of cyclophosphamide (Cytoxan) and high-dose immunosuppressive therapy with autologous stem cell transplantation on thymopoiesis, and [3] to describe the kinetics and breadth of T cell immune recovery in SSc patients treated with these interventions.

ELIGIBILITY:
Inclusion Criteria:

* Severe systemic sclerosis (SSc) as defined by the American College of Rheumatology (ACR);
* SSc, including extensive skin and internal organ involvement involving either the lungs or the kidneys, that threatens participant's life; and
* Willingness to use accepted methods of contraception for at least 15 months after starting study treatment.

Exclusion Criteria:

* Lung, heart, liver, or kidney impairment that would interfere with the study or compromise participant's survival;
* Active blood vessel dilation in the stomach (Active Gastric Antral Vascular Ectasia/GAVE, also known as "watermelon stomach"). Patients found to have this disorder at study screening can receive treatment outside the study and then be re-screened. For more information about this study criterion, refer to the study protocol.
* Previous treatment with cyclophosphamide, as defined by: a) prior IV cyclophosphamide administration for more than 6 months OR a total cumulative IV dose greater than 3 g/m^2; b) prior oral cyclophosphamide administration for more than 4 months, regardless of dose; or c) combination of prior oral and IV cyclophosphamide administration for more than 6 months, independent of dose.
* Steroid therapy at doses of greater than 10 mg/day, or more than 2 pulses for concurrent illnesses within prior 12 months;
* Unwillingness or inability to discontinue certain disease-modifying antirheumatic drugs (DMARDs) for the treatment of SSc;
* Presence of clinically significant rheumatic diseases other than scleroderma requiring significant immunosuppression;
* Any active uncontrolled infection that would interfere with high-dose therapy or pulse cyclophosphamide regimens:

  * Hepatitis B virus infected
  * Hepatitis C virus infected or
  * HIV infected.
* Blood abnormalities;
* Diagnosis of cancer within 2 years prior to study entry. Participants with adequately treated squamous cell skin cancer, basal cell carcinoma, and carcinoma in situ are not excluded.
* Other comorbid illnesses with an estimated life expectancy of less than 5 years;
* Defective formation of bone marrow cells (myelodysplasia);
* Uncontrolled hypertension;
* History of hypersensitivity to murine or Escherichia coli (e.g., E. coli) proteins; History of noncompliance with prior medical care;
* History of substance abuse within 5 years prior to study entry; or
* Pregnancy.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith M. Sullivan, MD, Study Chair — Duke University; Daniel E. Furst, MD, Study Chair — University of California, Los Angeles Rheumatology; Peter A. McSweeney, MD, Study Chair — Presbyterian/St. Luke's Medical Center:Rocky Mountain Cancer Center; Leslie J. Crofford, MD, Principal Investigator — University of Kentucky, Women's Health Program: Rheumatology; Maureen D. Mayes, MD, MPH, Principal Investigator — University of Texas - Houston Health Science Center; Richard A. Nash, MD, Principal Investigator — Fred Hutchinson Cancer Research
Locations (17):
- United States (15):
  - City of Hope National Medical Center, Duarte, California
  - UCLA Medical School, Los Angeles, California
  - University of Kentucky, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - University of Toledo Health Science Campus, Toledo, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas-Houston Medical School, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center (FHCRC), Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Dr. Markland Medical Professional Corporation, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share IPD in the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts. This archive is in support of the NIH mission to share data with the public. Data shared through ImmPort has been provided by NIH-funded programs, other research organizations and individual scientists ensuring these discoveries will be the foundation of future research.

REFERENCES:
- [Background] Nash RA, McSweeney PA, Crofford LJ, Abidi M, Chen CS, Godwin JD, Gooley TA, Holmberg L, Henstorf G, LeMaistre CF, Mayes MD, McDonagh KT, McLaughlin B, Molitor JA, Nelson JL, Shulman H, Storb R, Viganego F, Wener MH, Seibold JR, Sullivan KM, Furst DE. High-dose immunosuppressive therapy and autologous hematopoietic cell transplantation for severe systemic sclerosis: long-term follow-up of the US multicenter pilot study. Blood. 2007 Aug 15;110(4):1388-96. doi: 10.1182/blood-2007-02-072389. Epub 2007 Apr 23. PMID 17452515
- [Background] Sullivan KM, Shah A, Sarantopoulos S, Furst DE. Review: Hematopoietic Stem Cell Transplantation for Scleroderma: Effective Immunomodulatory Therapy for Patients With Pulmonary Involvement. Arthritis Rheumatol. 2016 Oct;68(10):2361-71. doi: 10.1002/art.39748. No abstract available. PMID 27213276
- [Result] Craciunescu OI, Steffey BA, Kelsey CR, Larrier NA, Paarz-Largay CJ, Prosnitz RG, Chao N, Chute J, Gasparetto C, Horwitz M, Long G, Rizzieri D, Sullivan KM. Renal shielding and dosimetry for patients with severe systemic sclerosis receiving immunoablation with total body irradiation in the scleroderma: cyclophosphamide or transplantation trial. Int J Radiat Oncol Biol Phys. 2011 Mar 15;79(4):1248-55. doi: 10.1016/j.ijrobp.2010.05.036. Epub 2010 Aug 26. PMID 20800376
- [Result] Hosing C, Nash R, McSweeney P, Mineishi S, Seibold J, Griffith LM, Shulman H, Goldmuntz E, Mayes M, Parikh CR, Crofford L, Keyes-Elstein L, Furst D, Steen V, Sullivan KM. Acute kidney injury in patients with systemic sclerosis participating in hematopoietic cell transplantation trials in the United States. Biol Blood Marrow Transplant. 2011 May;17(5):674-81. doi: 10.1016/j.bbmt.2010.08.003. Epub 2010 Aug 11. PMID 20708086
- [Result] Hung EW, Mayes MD, Sharif R, Assassi S, Machicao VI, Hosing C, St Clair EW, Furst DE, Khanna D, Forman S, Mineishi S, Phillips K, Seibold JR, Bredeson C, Csuka ME, Nash RA, Wener MH, Simms R, Ballen K, Leclercq S, Storek J, Goldmuntz E, Welch B, Keyes-Elstein L, Castina S, Crofford LJ, Mcsweeney P, Sullivan KM. Gastric antral vascular ectasia and its clinical correlates in patients with early diffuse systemic sclerosis in the SCOT trial. J Rheumatol. 2013 Apr;40(4):455-60. doi: 10.3899/jrheum.121087. Epub 2013 Feb 15. PMID 23418384
- [Result] Keever-Taylor CA, Heimfeld S, Steinmiller KC, Nash RA, Sullivan KM, Czarniecki CW, Granderson TC, Goldstein JS, Griffith LM. Manufacture of Autologous CD34+ Selected Grafts in the NIAID-Sponsored HALT-MS and SCOT Multicenter Clinical Trials for Autoimmune Diseases. Biol Blood Marrow Transplant. 2017 Sep;23(9):1463-1472. doi: 10.1016/j.bbmt.2017.05.018. Epub 2017 Jun 30. PMID 28602891
- [Result] Sullivan KM, Goldmuntz EA, Keyes-Elstein L, McSweeney PA, Pinckney A, Welch B, Mayes MD, Nash RA, Crofford LJ, Eggleston B, Castina S, Griffith LM, Goldstein JS, Wallace D, Craciunescu O, Khanna D, Folz RJ, Goldin J, St Clair EW, Seibold JR, Phillips K, Mineishi S, Simms RW, Ballen K, Wener MH, Georges GE, Heimfeld S, Hosing C, Forman S, Kafaja S, Silver RM, Griffing L, Storek J, LeClercq S, Brasington R, Csuka ME, Bredeson C, Keever-Taylor C, Domsic RT, Kahaleh MB, Medsger T, Furst DE; SCOT Study Investigators. Myeloablative Autologous Stem-Cell Transplantation for Severe Scleroderma. N Engl J Med. 2018 Jan 4;378(1):35-47. doi: 10.1056/nejmoa1703327. PMID 29298160
- [Result] Bellocchi C, Ying J, Goldmuntz EA, Keyes-Elstein L, Varga J, Hinchcliff ME, Lyons MA, McSweeney P, Furst DE, Nash R, Crofford LJ, Welch B, Goldin JG, Pinckney A, Mayes MD, Sullivan KM, Assassi S. Large-Scale Characterization of Systemic Sclerosis Serum Protein Profile: Comparison to Peripheral Blood Cell Transcriptome and Correlations With Skin/Lung Fibrosis. Arthritis Rheumatol. 2021 Apr;73(4):660-670. doi: 10.1002/art.41570. Epub 2021 Feb 28. PMID 33131208
- [Result] Keyes-Elstein L, Pinckney A, Goldmuntz E, Welch B, Franks JM, Martyanov V, Wood TA, Crofford L, Mayes M, McSweeney P, Nash R, Georges G, Csuka ME, Simms R, Furst D, Khanna D, Clair EWS, Whitfield ML, Sullivan KM. Clinical and Molecular Findings After Autologous Stem Cell Transplantation or Cyclophosphamide for Scleroderma: Handling Missing Longitudinal Data. Arthritis Care Res (Hoboken). 2023 Feb;75(2):307-316. doi: 10.1002/acr.24785. Epub 2022 Nov 16. PMID 34533286
- [Derived] Bruera S, Sidanmat H, Molony DA, Mayes MD, Suarez-Almazor ME, Krause K, Lopez-Olivo MA. Stem cell transplantation for systemic sclerosis. Cochrane Database Syst Rev. 2022 Jul 29;7(7):CD011819. doi: 10.1002/14651858.CD011819.pub2. PMID 35904231
- [Derived] Shah A, Storek J, Woolson R, Pinckney A, Keyes-Elstein L, Wallace PK, Sempowski GD, McSweeney P, Mayes MD, Crofford L, Csuka ME, Phillips K, Khanna D, Simms R, Ballen K, LeClercq S, Clair WS, Nixon AB, Nash R, Wener M, Brasington R, Silver R, Griffith LM, Furst DE, Goldmuntz E, Sullivan KM. Lymphocyte subset abnormalities in early severe scleroderma favor a Th2 phenotype and are not altered by prior immunosuppressive therapy. Rheumatology (Oxford). 2022 Oct 6;61(10):4155-4162. doi: 10.1093/rheumatology/keac015. PMID 35108379
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Scleroderma: Cyclophosphamide or Transplantation (SCOT) Study — http://www.sclerodermatrial.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- mHSCT: Participants were administered granulocyte colony stimulating factor (G-CSF) and had hematopoietic stem cells removed from their blood. They then underwent high-dose immunosuppressive therapy using a conditioning regimen of total body irradiation (800 cGy given over 2 days with lung and kidney shielding limiting exposure to 200cGy), cyclophosphamide (60 mg/kg/day for 2 days), IV Methylprednisolone (1 mg/kg/day for 3 days), and equine antithymocyte globulin (ATGAM) (15 mg/kg/day for 3 days). Purified autologous stem cell were infused at a dose of >2.5x106 CD34+ cells/kg. After transplantation, participants received additional doses of IV Methylprednisolone (1 mg/kg/day for 3 days) and ATGAM (15 mg/kg/day for 3 days.)
- Cyclophosphamide: Participants received 12 monthly pulses of high-dose intravenous cyclophosphamide (an initial dose of 500 mg/m^2, followed by 11 doses of 750 mg/m^2).
Period: Overall Study
Arm/Group | mHSCT | Cyclophosphamide
Started | 36 | 39
Completed | 27 (Completed 72 mo, 54 mo after failure, or at least 54 mo at study end (last patient's 54 mo visit)) | 19 (Completed 72 mo, 54 mo after failure, or at least 54 mo at study end (last patient's 54 mo visit))
Not Completed | 9 | 20
Not completed — Death | 3 | 11
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Breast Cancer | 1 | 0
Not completed — Subject decision after endpoint failure | 0 | 1
Not completed — Ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized intent to treat
Groups:
- Total: Total of all reporting groups
Arm/Group | mHSCT | Cyclophosphamide | Total
Number analyzed (Participants) | 36 | 39 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 38 | 73
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (10.90) | 46.9 (10.43) | 45.9 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 29 | 48
  Male | 17 | 10 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 32 | 34 | 66
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 29 | 31 | 60
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 2 | 3
  United States | 35 | 37 | 72
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — HAQ-DI is a self-reported questionnaire of functionality that includes questions in 8 domains (dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities). The final score ranges from 0 to 3, where a higher HAQ-DI score indicates a worse outcome.
  units on a scale | 1.2 (0.65) | 1.4 (0.86) | 1.3 (0.77)
Short Form 36 Health Survey (SF-36) [Mean (Standard Deviation); unit: units on a scale] — The SF-36 measures health-related quality of life. It has 36 items and 2 component scores, the Physical Component Score and the Mental Component Score. Each component was transformed into a 0-100 scale (higher numbers indicate greater quality of life) and normalized to have a mean of 50 and standard deviation of 10 for the 1998 general US population.
  units on a scale
    Physical Component Score | 29.5 (9.20) | 28.9 (9.46) | 29.2 (9.27)
    Mental Component Score | 44.7 (10.70) | 44.6 (9.86) | 44.6 (10.21)
Diffusion in Liters of Carbon Monoxide (DLCO) (Percent-Predicted) [Mean (Standard Deviation); unit: Percent predicted] — Diffusion in liters of carbon monoxide (DLCO) is a measure of lung function. Predicted values for DLCO were computed using the Crapo Morris equations and adjusted per the Cotes formula for anemia, if a participant's hemoglobin was <13 or >17 gm/dL, and altitude (Calgary site only).
  Percent predicted | 53.9 (7.63) | 52.7 (8.19) | 53.3 (7.90)
Forced Vital Capacity (FVC) (Percent-Predicted) [Mean (Standard Deviation); unit: percent predicted] — Forced Vital Capacity (FVC) is the amount of air that can be forcibly exhaled after a full breath and is a measure of lung function. Predicted FVC was based on institutional standards.
  percent predicted | 74.5 (14.77) | 73.8 (16.98) | 74.2 (15.86)
Modified Rodnan Skin Score (mRSS) [Mean (Standard Deviation); unit: units on a scale] — The Modified Rodnan Skin Score (mRSS) is a measure of skin thickness. Skin thickness in 17 anatomic areas was rated on a 0-3 scale and scores are summed to obtain the mRSS (range from 0 - 51), with higher mRSS scores indicating worse disease activity.
  units on a scale | 28.5 (8.72) | 30.8 (10.55) | 29.7 (9.72)
Disease-Modifying Anti-Rheumatic Drug (DMARD) Use Within 6 Months of Randomization [Count of Participants; unit: Participants] — Use of any disease-modifying antirheumatic drugs (DMARDs) within six months prior to randomization. DMARDS can include, but are not limited to, methotrexate, cyclophosphamide, azathioprine, leflunomide, mycophenolate mofetil, D-penicillamine, tacrolimus, cyclosporine, prednisone >10 mg, and TNF-blockers.
  Participants | 26 | 25 | 51
Disease-Modifying Anti-Rheumatic Drug (DMARD) Use [Count of Participants; unit: Participants] — Any use of disease-modifying antirheumatic drugs (DMARDs) prior to randomization. DMARDS can include, but are not limited to, methotrexate, cyclophosphamide, azathioprine, leflunomide, mycophenolate mofetil, D-penicillamine, tacrolimus, cyclosporine, prednisone >10 mg, and TNF-blockers.
  Participants | 27 | 32 | 59

OUTCOME MEASURES:

1. Primary Outcome: Global Rank Composite Score (GRCS) (Month 54, ITT)
Description: The GRCS is an analytic tool that accounts for multiple disease manifestations simultaneously. It does not measure clinical disease activity or severity but reflects how participants compared to one another based on a hierarchy of ordered outcomes: death, event-free survival (EFS), forced vital capacity (FVC), Health Assessment Questionnaire - Disability Index (HAQ-DI), and Modified Rodnan Skin Score (mRSS). Participants alive ranked higher than those who died; those who survived event-free ranked higher than EFS failures. EFS failure included death, respiratory failure (decrease from baseline of >30% in DLCO % predicted or >20% in FVC % predicted ), renal failure (chronic dialysis > 6 month or renal transplant), or cardiac failure (clinical congestive heart failure or left ventricular ejection fraction <30%). The lowest 3 GRCS components are ordinal; improvement, stability, or worsening from baseline (±10% change in FVC % predicted, ±0.4 change in HAQ-DI, ±25% change in mRSS).
Time Frame: 54 Months Post-Randomization
Population: Intention to treat (ITT). The ITT population includes all randomized participants.
Measure: Median (Full Range); unit: Sum of subject-pair comparison scores
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 36 | 39
Sum of subject-pair comparison scores | 17.0 [-58 to 52] | -6.0 [-58 to 52]
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.013, Wilcoxon (Mann-Whitney) — A Data and Safety Monitoring Board reviewed 4 pre-specified futility analyses that included an ability to stop for efficacy with p<0.0001, leaving alpha equal to 0.0496 for the primary ITT analysis of the GRCS at 54 months post-randomization

2. Secondary Outcome: Global Rank Composite Score (GRCS) (Month 54, PP)
Description: as for outcome 1
Time Frame: 54 Months Post-Randomization
Population: Per-protocol (PP). The PP population is defined as those participants who completed the assigned treatment protocol: undergoing autologous CD34-selected hematopoietic progenitor cell transplantation in the mHSCT arm, or receiving at least 9 of 12 planned doses in the cyclophosphamide arm.
Measure: Median (Full Range); unit: Sum of subject-pair comparison scores
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 33 | 34
Sum of subject-pair comparison scores | 16 [-56 to 46] | -11.0 [-56 to 46]
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Global Rank Composite Score (GRCS) (Month 48, ITT)
Description: as for outcome 1
Time Frame: 48 Months Post-Randomization
Population: Intention to treat (ITT). The ITT population includes all randomized participants.
Measure: Median (Full Range); unit: Sum of subject-pair comparison scores
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 36 | 39
Sum of subject-pair comparison scores | 20.0 [-58 to 55] | -8.0 [-58 to 55]
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.008, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Global Rank Composite Score (GRCS) (Month 48, PP)
Description: as for outcome 1
Time Frame: 48 Months Post-Randomization
Population: as for outcome 2
Measure: Median (Full Range); unit: Sum of subject-pair comparison scores
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 33 | 34
Sum of subject-pair comparison scores | 17.0 [-56 to 49] | -13.0 [-56 to 49]
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Event-Free Survival (EFS) (Month 54, ITT)
Description: Event-free survival (EFS) is defined as survival without significant organ damage or death. EFS failure includes any one of the following: death, respiratory failure (decrease from baseline of >30% in diffusion in liters of carbon monoxide (DLCO) % predicted or >20% in forced vital capacity (FVC) % predicted, documented on at least 2 successive occasions at least 1 month apart), renal failure (requiring chronic dialysis > 6 months or transplantation), or the occurrence of cardiomyopathy (clinical congestive heart failure or left ventricular ejection fraction <30%, documented on at least 2 successive occasions at least 1 month apart). EFS failures include participants who failed any component of the EFS definition between randomization and Month 54 post-randomization.
Time Frame: 54 Months Post-Randomization
Population: Intention to treat (ITT). The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 36 | 39
Participants
  EFS Failure | 10 | 20
  Survived Event Free | 26 | 19
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Treatment arm comparisons of EFS at Month 54; Test type: Superiority; p = 0.059, Fisher Exact
Statistical Analysis 2: Comparison: mHSCT vs Cyclophosphamide; Treatment arm comparisons of Kaplan-Meier curves for EFS through Month 72; Test type: Superiority; p = 0.06, Log Rank

6. Secondary Outcome: Event-Free Survival (EFS) (Month 54, PP)
Description: Event-free survival (EFS) is defined as survival without significant organ damage or death. EFS failure includes any one of the following: death, respiratory failure (decrease from baseline of >30% in DLCO % predicted or >20% in FVC % predicted, documented on at least 2 successive occasions at least 1 month apart), renal failure (requiring chronic dialysis > 6 months or transplantation), or the occurrence of cardiomyopathy (clinical congestive heart failure or left ventricular ejection fraction <30%, documented on at least 2 successive occasions at least 1 month apart). EFS failures include participants who failed any component of the EFS definition between randomization and Month 54 post-randomization.
Time Frame: 54 Months Post-Randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 33 | 34
Participants
  EFS Failure | 7 | 17
  Survived Event Free | 26 | 17
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Treatment arm comparisons of EFS at Month 54; Test type: Superiority; p = 0.021, Fisher Exact
Statistical Analysis 2: Comparison: mHSCT vs Cyclophosphamide; Treatment arm comparisons of Kaplan-Meier curves for EFS through Month 72; Test type: Superiority; p = 0.03, Log Rank

7. Secondary Outcome: Event-Free Survival (EFS) (Month 48, ITT)
Description: Event-free survival (EFS) is defined as survival without significant organ damage or death. EFS failure includes any one of the following: death, respiratory failure (decrease from baseline of >30% in DLCO % predicted or >20% in FVC % predicted, documented on at least 2 successive occasions at least 1 month apart), renal failure (requiring chronic dialysis > 6 months or transplantation), or the occurrence of cardiomyopathy (clinical congestive heart failure or left ventricular ejection fraction <30%, documented on at least 2 successive occasions at least 1 month apart). EFS failures include participants who failed any component of the EFS definition between randomization and Month 48 post-randomization.
Time Frame: 48 Months Post-Randomization
Population: Intention to treat (ITT). The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 36 | 39
Participants
  EFS Failure | 10 | 20
  Survived Event Free | 26 | 19
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.059, Fisher Exact

8. Secondary Outcome: Event-Free Survival (EFS) (Month 48, PP)
Description: as for outcome 7
Time Frame: 48 Months Post-Randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 33 | 34
Participants
  EFS Failure | 7 | 17
  Survived Event Free | 26 | 17
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.021, Fisher Exact

9. Secondary Outcome: Treatment-Related Mortality (Month 54, ITT)
Description: Death, occurring at any time between randomization and Month 54 post-randomization, which is possibly, probably, or definitely resulting from treatment given in the study.
Time Frame: 54 Months Post-Randomization
Population: Intention to treat (ITT). The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 36 | 39
Participants | 1 | 0
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.48, Fisher Exact

10. Secondary Outcome: Treatment-Related Mortality (Month 54, PP)
Description: as for outcome 9
Time Frame: 54 Months Post-Randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 33 | 34
Participants | 1 | 0
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.49, Fisher Exact

11. Secondary Outcome: Treatment-Related Mortality (Month 48, ITT)
Description: Death, occurring at any time between randomization and Month 48 post-randomization, which is possibly, probably, or definitely resulting from treatment given in the study.
Time Frame: 48 Months Post-Randomization
Population: Intention to treat (ITT). The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 36 | 39
Participants | 1 | 0
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.48, Fisher Exact

12. Secondary Outcome: Treatment-Related Mortality (Month 48, PP)
Description: as for outcome 11
Time Frame: 48 Months Post-Randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 33 | 34
Participants | 1 | 0
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.49, Fisher Exact

13. Secondary Outcome: All-Cause Mortality (Month 54, ITT)
Description: Any death, regardless of relationship to treatment, between randomization and Month 54 post-randomization.
Time Frame: 54 Months Post-Randomization
Population: Intention to treat (ITT). The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 36 | 39
Participants | 6 | 11
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Treatment arm comparisons of overall survival at Month 54; Test type: Superiority; p = 0.28, Fisher Exact
Statistical Analysis 2: Comparison: mHSCT vs Cyclophosphamide; Treatment arm comparisons of Kaplan-Meier curves for overall survival through Month 72; Test type: Superiority; p = 0.05, Log Rank

14. Secondary Outcome: All-Cause Mortality (Month 54, PP)
Description: Any death, regardless of relationship to treatment, between randomization and Month 54 post-randomization.
Time Frame: 54 Months Post-Randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 33 | 34
Participants | 3 | 8
Statistical Analysis 1: Comparison: mHSCT; Treatment arm comparisons of overall survival at Month 54; Test type: Superiority; p = 0.19, Fisher Exact
Statistical Analysis 2: Comparison: mHSCT vs Cyclophosphamide; Treatment arm comparisons of Kaplan-Meier curves for overall survival through Month 72; Test type: Superiority; p = 0.02, Log Rank

15. Secondary Outcome: All-Cause Mortality (Month 48, ITT)
Description: Any death, regardless of relationship to treatment, between randomization and Month 48 post-randomization.
Time Frame: 48 Months Post-Randomization
Population: Intention to treat (ITT). The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 36 | 39
Participants | 6 | 11
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.28, Fisher Exact

16. Secondary Outcome: All-Cause Mortality (Month 48, PP)
Description: Any death, regardless of relationship to treatment, between randomization and Month 48 post-randomization.
Time Frame: 48 Months Post-Randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 33 | 34
Participants | 3 | 8
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.19, Fisher Exact

17. Secondary Outcome: Change From Baseline to Month 54 in Health Assessment Questionnaire - Disability Index (HAQ-DI) (ITT)
Description: HAQ-DI is a self-reported questionnaire of functionality that includes questions in 8 domains (dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities). The final score ranges from 0 to 3, where a higher HAQ-DI score indicates a worse outcome. Analysis was based on an ordinal response variable, defined as follows: a decrease of >0.4 from baseline in the HAQ-DI score was considered disease improvement, an increase of >0.4 was considered disease worsening, and any change less than 0.4 was considered "no change." Data for participants without a Month 54 assessment was imputed using a last observation carried forward approach; improvement/worsening was assessed at each participant's last available study visit that occurred prior to or at Month 54, without confirmation at the next visit.
Time Frame: 54 Months Post-Randomization
Population: Intention to treat (ITT). The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Groups:
- mHSCT- EFS Survivor: Subjects in the mHSCT group who met the event-free survival (EFS) endpoint, defined as survival without significant organ damage or death.
- Cyclophosphamide-EFS Survivor: Subjects in the Cyclophosphamide group who met the event-free survival (EFS) endpoint, defined as survival without significant organ damage or death.
- mHSCT- EFS Failure: Subjects in the mHSCT group who failed the event-free survival (EFS) endpoint, defined as survival without significant organ damage or death.
- Cyclophosphamide- EFS Failure: Subjects in the Cyclophosphamide group who failed the event-free survival (EFS) endpoint, defined as survival without significant organ damage or death.
Arm/Group | mHSCT- EFS Survivor | Cyclophosphamide-EFS Survivor | mHSCT- EFS Failure | Cyclophosphamide- EFS Failure
Number analyzed (Participants) | 26 | 19 | 10 | 20
Participants
  Improvement | 17 | 6 | 2 | 0
  No Change | 8 | 11 | 5 | 11
  Worsening | 1 | 2 | 3 | 9
Statistical Analysis 1: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; This analysis is not stratified. EFS survivors and failures are pooled within each treatment arm; Test type: Superiority; p < 0.001, Kruskal-Wallis; Computed as Mantel Haenszel Chi Square using modified ridit scores
Statistical Analysis 2: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; This analysis is stratified by EFS status; Test type: Superiority; p = 0.01, Wilcoxon (Mann-Whitney); Van Elteren extension of the Wilcoxon Rank Sum

18. Secondary Outcome: Change From Baseline to Month 54 in Health Assessment Questionnaire - Disability Index (HAQ-DI) (PP)
Description: as for outcome 17
Time Frame: 54 Months Post-Randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT- EFS Survivor | Cyclophosphamide-EFS Survivor | mHSCT- EFS Failure | Cyclophosphamide- EFS Failure
Number analyzed (Participants) | 26 | 17 | 7 | 17
Participants
  Improvement | 17 | 6 | 2 | 0
  No Change | 8 | 10 | 5 | 9
  Worsening | 1 | 1 | 0 | 8
Statistical Analysis 1: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; This analysis is not stratified. EFS survivors and failures are pooled within each treatment arm; Test type: Superiority; p < 0.001, Kruskal-Wallis; Computed as Mantel Haenszel Chi Square using modified ridit scores
Statistical Analysis 2: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; This analysis is stratified by EFS status; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney); Van Elteren extension of the Wilcoxon Rank Sum

19. Secondary Outcome: Change From Baseline to Month 54 in Short Form 36 Health Survey (SF-36) (ITT)
Description: The SF-36 measures health-related quality of life. It has 36 items and 2 component scores, the Physical Component Score and the Mental Component Score. Each component was transformed into a 0-100 scale (higher numbers indicate greater quality of life) and normalized to have a mean of 50 and standard deviation of 10 for the 1998 general US population. Analysis was based on ordinal response, defined as follows for each component: a >= 10 point increase indicated disease improvement, a >= 10 point decrease indicated disease worsening, and a change <10 points indicated "no change". Data for participants without a Month 54 assessment was imputed using a last observation carried forward approach; improvement/worsening was assessed at each participant's last available study visit that occurred prior to or at Month 54, without confirmation at the next visit.
Time Frame: 54 Months Post-Randomization
Population: Intention to treat (ITT). The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT- EFS Survivor | Cyclophosphamide-EFS Survivor | mHSCT- EFS Failure | Cyclophosphamide- EFS Failure
Number analyzed (Participants) | 26 | 19 | 10 | 20
Participants
  Physical Component Score: Improvement | 19 | 6 | 1 | 0
  Physical Component Score: No Change | 6 | 9 | 6 | 16
  Physical Component Score: Worsening | 1 | 4 | 3 | 4
  Mental Component Score: Improvement | 10 | 2 | 1 | 1
  Mental Component Score: No Change | 12 | 12 | 5 | 12
  Mental Component Score: Worsening | 4 | 5 | 4 | 7
Statistical Analysis 1: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; Physical Component Score. This analysis is not stratified. EFS survivors and failures are pooled within each treatment arm; Test type: Superiority; p = 0.001, Kruskal-Wallis; Computed as Mantel Haenszel Chi Square using modified ridit scores
Statistical Analysis 2: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; Physical Component Score. This analysis is stratified by EFS status; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney); Van Elteren extension of the Wilcoxon Rank Sum
Statistical Analysis 3: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; Mental Component Score. This analysis is not stratified. EFS survivors and failures are pooled within each treatment arm; Test type: Superiority; p = 0.05, Kruskal-Wallis; Computed as Mantel Haenszel Chi Square using modified ridit scores
Statistical Analysis 4: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; Mental Component Score. This analysis is stratified by EFS status; Test type: Superiority; p = 0.1, Wilcoxon (Mann-Whitney); Van Elteren extension of the Wilcoxon Rank Sum

20. Secondary Outcome: Change From Baseline to Month 54 in Short Form 36 Health Survey (SF-36) (PP)
Description: as for outcome 19
Time Frame: 54 Months Post-Randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT- EFS Survivor | Cyclophosphamide-EFS Survivor | mHSCT- EFS Failure | Cyclophosphamide- EFS Failure
Number analyzed (Participants) | 26 | 17 | 7 | 17
Participants
  Physical Component Score: Improvement | 19 | 6 | 1 | 0
  Physical Component Score: No Change | 6 | 9 | 6 | 14
  Physical Component Score: Worsening | 1 | 2 | 0 | 3
  Mental Component Score: Improvement | 10 | 2 | 1 | 1
  Mental Component Score: No Change | 12 | 12 | 5 | 10
  Mental Component Score: Worsening | 4 | 3 | 1 | 6
Statistical Analysis 1: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p < 0.001, Kruskal-Wallis; Computed as Mantel Haenszel Chi Square using modified ridit scores
Statistical Analysis 2: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; Physical Component Score. This analysis is stratified by EFS status; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney); Van Elteren extension of the Wilcoxon Rank Sum
Statistical Analysis 3: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; [analysis description as in outcome 19, analysis 3]; Test type: Superiority; p = 0.02, Kruskal-Wallis; Computed as Mantel Haenszel Chi Square using modified ridit scores
Statistical Analysis 4: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; Mental Component Score. This analysis is stratified by EFS status; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney); Van Elteren extension of the Wilcoxon Rank Sum

21. Secondary Outcome: Change From Baseline to Month 54 in Diffusion in Liters of Carbon Monoxide (DLCO) (ITT)
Description: Diffusion in liters of carbon monoxide (DLCO) is a measure of lung function. Predicted values for DLCO were computed using the Crapo Morris equations and adjusted per the Cotes formula for anemia, if a participant's hemoglobin was <13 or >17 gm/dL, and altitude (Calgary site only). Analysis was based on an ordinal response variable, defined as follows: an increase from baseline of >15% in DLCO % Predicted indicated disease improvement, a decrease of >15% indicated disease worsening, and a change of <=15% was considered "no change". Data for participants without a Month 54 assessment was imputed using a last observation carried forward approach; improvement/worsening was assessed at each participant's last available study visit that occurred prior to or at Month 54, without confirmation at the next visit.
Time Frame: 54 Months Post-Randomization
Population: Intention to treat (ITT). The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT- EFS Survivor | Cyclophosphamide-EFS Survivor | mHSCT- EFS Failure | Cyclophosphamide- EFS Failure
Number analyzed (Participants) | 26 | 19 | 10 | 20
Participants
  Improvement | 4 | 5 | 0 | 0
  No Change | 19 | 8 | 0 | 2
  Worsening | 3 | 6 | 10 | 18
Statistical Analysis 1: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; This analysis is not stratified. EFS survivors and failures are pooled within each treatment arm; Test type: Superiority; p = 0.08, Kruskal-Wallis; Computed as Mantel Haenszel Chi Square using modified ridit scores
Statistical Analysis 2: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; This analysis is stratified by EFS status; Test type: Superiority; p = 0.9, Wilcoxon (Mann-Whitney); Van Elteren extension of the Wilcoxon Rank Sum

22. Secondary Outcome: Change From Baseline to Month 54 in Diffusion in Liters of Carbon Monoxide (DLCO) (PP)
Description: as for outcome 21
Time Frame: 54 Months Post-Randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT- EFS Survivor | Cyclophosphamide-EFS Survivor | mHSCT- EFS Failure | Cyclophosphamide- EFS Failure
Number analyzed (Participants) | 26 | 17 | 7 | 17
Participants
  Improvement | 4 | 5 | 0 | 0
  No Change | 19 | 8 | 0 | 2
  Worsening | 3 | 4 | 7 | 15
Statistical Analysis 1: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; This analysis is not stratified. EFS survivors and failures are pooled within each treatment arm; Test type: Superiority; p = 0.1, Kruskal-Wallis; Computed as Mantel Haenszel Chi Square using modified ridit scores
Statistical Analysis 2: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; This analysis is stratified by EFS status; Test type: Superiority; p = 0.6, Wilcoxon (Mann-Whitney); Van Elteren extension of the Wilcoxon Rank Sum

23. Secondary Outcome: Change From Baseline to Month 54 in Forced Vital Capacity (FVC) (ITT)
Description: Forced Vital Capacity (FVC) is the amount of air that can be forcibly exhaled after a full breath and is a measure of lung function. Predicted FVC was based on institutional standards. Analysis was based on an ordinal response variable, defined as follows: an increase from baseline of >10% in FVC % Predicted indicated disease improvement, a decrease of >10% indicated disease worsening, and a change of <=10% was considered "no change". Data for participants without a Month 54 assessment was imputed using a last observation carried forward approach; improvement/worsening was assessed at each participant's last available study visit that occurred prior to or at Month 54, without confirmation at the next visit.
Time Frame: 54 Months Post-Randomization
Population: Intention to treat (ITT). The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT- EFS Survivor | Cyclophosphamide-EFS Survivor | mHSCT- EFS Failure | Cyclophosphamide- EFS Failure
Number analyzed (Participants) | 26 | 19 | 10 | 20
Participants
  Improvement | 12 | 7 | 0 | 1
  No Change | 13 | 8 | 2 | 2
  Worsening | 1 | 4 | 8 | 17
Statistical Analysis 1: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; This analysis is not stratified. EFS survivors and failures are pooled within each treatment arm; Test type: Superiority; p = 0.02, Kruskal-Wallis; Computed as Mantel Haenszel Chi Square using modified ridit scores
Statistical Analysis 2: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; This analysis is stratified by EFS status; Test type: Superiority; p = 0.3, Wilcoxon (Mann-Whitney); Van Elteren extension of the Wilcoxon Rank Sum

24. Secondary Outcome: Change From Baseline to Month 54 in Forced Vital Capacity (FVC) (PP)
Description: as for outcome 23
Time Frame: 54 Months Post-Randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT- EFS Survivor | Cyclophosphamide-EFS Survivor | mHSCT- EFS Failure | Cyclophosphamide- EFS Failure
Number analyzed (Participants) | 26 | 17 | 7 | 17
Participants
  Improvement | 12 | 7 | 0 | 1
  No Change | 13 | 8 | 2 | 2
  Worsening | 1 | 2 | 5 | 14
Statistical Analysis 1: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; This analysis is not stratified. EFS survivors and failures are pooled within each treatment arm; Test type: Superiority; p = 0.03, Kruskal-Wallis; Computed as Mantel Haenszel Chi Square using modified ridit scores
Statistical Analysis 2: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; This analysis is stratified by EFS status; Test type: Superiority; p = 0.5, Wilcoxon (Mann-Whitney); Van Elteren extension of the Wilcoxon Rank Sum

25. Secondary Outcome: Change From Baseline to Month 54 in Modified Rodnan Skin Score (mRSS) (ITT)
Description: The Modified Rodnan Skin Score (mRSS) is a measure of skin thickness. Skin thickness in 17 anatomic areas was rated on a 0-3 scale and scores are summed to obtain the mRSS (range from 0 - 51), with higher mRSS scores indicating worse disease activity. Analysis was based on an ordinal response variable, defined as follows: if the baseline mRSS was <=20, a decrease >=5 points from baseline indicated disease improvement and an increase >= 5 points indicated disease worsening; if the baseline mRSS was >20, then a decrease of >25% indicated disease improvement and an increase of >25% indicated disease worsening. Participants who do not meet the disease criteria outlined above were considered "no change". Data for participants without a Month 54 assessment was imputed using a last observation carried forward approach; improvement/worsening was assessed at each participant's last available study visit that occurred prior to or at Month 54, without confirmation at the next visit.
Time Frame: 54 Months Post-Randomization
Population: Intention to treat (ITT). The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT- EFS Survivor | Cyclophosphamide-EFS Survivor | mHSCT- EFS Failure | Cyclophosphamide- EFS Failure
Number analyzed (Participants) | 26 | 19 | 10 | 20
Participants
  Improvement | 26 | 14 | 5 | 5
  No Change | 0 | 3 | 1 | 10
  Worsening | 0 | 2 | 4 | 5
Statistical Analysis 1: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; This analysis is not stratified. EFS survivors and failures are pooled within each treatment arm; Test type: Superiority; p = 0.002, Kruskal-Wallis; Computed as Mantel Haenszel Chi Square using modified ridit scores
Statistical Analysis 2: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; This analysis is stratified by EFS status; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney); Van Elteren extension of the Wilcoxon Rank Sum

26. Secondary Outcome: Change From Baseline to Month 54 in Modified Rodnan Skin Score (mRSS) (PP)
Description: as for outcome 25
Time Frame: 54 Months Post-Randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT- EFS Survivor | Cyclophosphamide-EFS Survivor | mHSCT- EFS Failure | Cyclophosphamide- EFS Failure
Number analyzed (Participants) | 26 | 17 | 7 | 17
Participants
  Improvement | 26 | 14 | 5 | 5
  No Change | 0 | 3 | 1 | 10
  Worsening | 0 | 0 | 1 | 2
Statistical Analysis 1: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; This analysis is not stratified. EFS survivors and failures are pooled within each treatment arm; Test type: Superiority; p < 0.001, Kruskal-Wallis; Computed as Mantel Haenszel Chi Square using modified ridit scores
Statistical Analysis 2: Comparison: mHSCT- EFS Survivor vs Cyclophosphamide-EFS Survivor vs mHSCT- EFS Failure vs Cyclophosphamide- EFS Failure; This analysis is stratified by EFS status; Test type: Superiority; p = 0.01, Wilcoxon (Mann-Whitney); Van Elteren extension of the Wilcoxon Rank Sum

27. Secondary Outcome: New or Worsening Arrhythmias, Congestive Heart Failure, or Pericardial Effusion (ITT)
Description: Any events that met the criteria outlined below or were reported as adverse events between randomization and Month 54 post-randomization are summarized. 1) Development of new or worsening arrhythmias that require medical treatment for >= 3 months or require ablative therapy or pacemaker insertion. (Note that for a participant who has medically controlled arrhythmia at randomization, worsening was defined as breakthrough episodes severe enough to prompt change in medication, an increase in the dose of a medication, or addition of a new medication to maintain control of the arrhythmia.) 2) Congestive heart failure (CHF) requiring clinical treatment for >= 3 months develops. 3) Clinically significant pericardial effusion (excess fluid around the heart) that required pericardial window.
Time Frame: 54 Months Post-Randomization
Population: Intention to treat (ITT). The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 36 | 39
Participants
  Development of new or worsening arrhythmias | 6 | 4
  CHF requiring clinical treatment | 0 | 4
  Clinically significant pericardial effusion | 2 | 1
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Development of new or worsening arrhythmias; Test type: Superiority; p = 0.42, Chi-squared
Statistical Analysis 2: Comparison: mHSCT vs Cyclophosphamide; CHF requiring clinical treatment; Test type: Superiority; p = 0.048, Chi-squared
Statistical Analysis 3: Comparison: mHSCT vs Cyclophosphamide; Clinically significant pericardial effusion; Test type: Superiority; p = 0.51, Chi-squared

28. Secondary Outcome: New or Worsening Arrhythmias, Congestive Heart Failure, or Pericardial Effusion (PP)
Description: Any events that met the criteria outlined below or were reported as adverse events between randomization and Month 54 post-randomization are summarized. 1) Development of new or worsening arrhythmias that require medical treatment for >= 3 months or require ablative therapy or pacemaker insertion. (Note that for a participant who has medically controlled arrhythmia at randomization, worsening will be defined as breakthrough episodes severe enough to prompt change in medication, an increase in the dose of a medication or addition of a new medication to maintain control of the arrhythmia.) 2) Congestive heart failure (CHF) requiring clinical treatment for >= 3 months develops. 3) Clinically significant pericardial effusion (excess fluid around the heart) that required pericardial window.
Time Frame: 54 Months Post-Randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 33 | 34
Participants
  Development of new or worsening arrhythmias | 6 | 4
  CHF requiring clinical treatment | 0 | 4
  Clinically significant pericardial effusion | 2 | 0
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Development of new or worsening arrhythmias; Test type: Superiority; p = 0.46, Chi-squared
Statistical Analysis 2: Comparison: mHSCT vs Cyclophosphamide; CHF requiring clinical treatment; Test type: Superiority; p = 0.042, Chi-squared
Statistical Analysis 3: Comparison: mHSCT vs Cyclophosphamide; Clinically significant pericardial effusion; Test type: Superiority; p = 0.15, Chi-squared

29. Secondary Outcome: New or Worsening Pulmonary Hypertension (ITT)
Description: Any pulmonary arterial hypertension (PAH) events that occurred between randomization and Month 54 post-randomization were summarized. Development of PAH occurred if the participant met the following criteria, where the measurement value(s) could not be explained by other causes such as congestive heart failure or pulmonary emboli: 1) a post-baseline peak systolic pulmonary artery pressure > 55 mmHg by echocardiogram or 2) a mean pulmonary artery pressure > 30 mmHg at rest measured by right heart catheterization. If the post-baseline peak systolic pulmonary artery pressure was between 40 to 55 mmHg by echocardiogram, a right heart catheterization was done to confirm a diagnosis of pulmonary artery hypertension. The endpoint was met if the mean pulmonary artery pressure was > 30 mmHg at rest by right heart catheterization. Additionally, any adverse event reported as PAH was included in the analysis.
Time Frame: 54 Months Post-Randomization
Population: Intention to treat (ITT). The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 36 | 39
Participants | 0 | 5
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.026, Chi-squared

30. Secondary Outcome: New or Worsening Pulmonary Hypertension (PP)
Description: Any pulmonary arterial hypertension (PAH) events that occurred between randomization and Month 54 post-randomization were summarized. Development of PAH occurred if the participant met the following criteria, where the measurement value(s) could not be explained by other causes such as congestive heart failure or pulmonary emboli: 1) a post-baseline peak systolic pulmonary artery pressure > 55 mmHg by echocardiogram or 2) a mean pulmonary artery pressure > 30 mmHg at rest measured by right heart catheterization. If the post-baseline peak systolic pulmonary artery pressure was between 40 to 55 mmHg by echocardiogram, a right heart catheterization would be done to confirm a diagnosis of pulmonary artery hypertension. The endpoint was met if the mean pulmonary artery pressure was > 30 mmHg at rest by right heart catheterization. Additionally, any adverse event reported as PAH was included in the analysis.
Time Frame: 54 Months Post-Randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 33 | 34
Participants | 0 | 5
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.022, Chi-squared

31. Secondary Outcome: Occurrence of Scleroderma Renal Crisis (ITT)
Description: Documented scleroderma renal crisis (hypertensive or non-hypertensive) occurring from randomization to Month 54 post-randomization was summarized. A hypertensive scleroderma renal crisis occurred if a participant obtained both of the following: New-onset hypertension, defined as systolic blood pressure (SBP) >= 140 mmHg, diastolic blood pressure (DBP) >= 90 mmHg, a rise in SBP >= 30 mmHg compared to baseline, or a rise in DBP >= 20 mmHg compared to baseline, and one of the following features: 1) increase of >= 50 % above baseline in serum creatinine, 2) proteinuria (>= 2+ by dipstick confirmed by protein:creatinine ratio > 2.5), 3) hematuria (>= 2+ by dipstick or > 10 RBCs/HPF, without menstruation), 4) thrombocytopenia (< 100,000 plts/mm3), or 5) hemolysis (determined by blood smear or increased reticulocyte count). Additionally, any adverse event reported as a scleroderma renal crisis was included in the analysis.
Time Frame: 54 Months Post-Randomization
Population: Intention to treat (ITT). The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 36 | 39
Participants | 2 | 3
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.71, Chi-squared

32. Secondary Outcome: Occurrence of Scleroderma Renal Crisis (PP)
Description: as for outcome 31
Time Frame: 54 Months Post-Randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 33 | 34
Participants | 0 | 1
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.32, Chi-squared

33. Secondary Outcome: Documented Myositis (ITT)
Description: Number of participants who experienced any event of myositis that occurred from randomization to Month 54 post-randomization. Documented myositis occurred if the participant had 1) elevated creatine phosphokinase (CPK), electromyography, and/or biopsy and 2) required > 30 mg per day prednisone for over 1 month or another therapy such as methotrexate (MTX) for treatment of myositis. Additionally, any adverse event reported as myositis was included in the analysis.
Time Frame: 54 Months Post-Randomization
Population: Intention to treat (ITT). The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 36 | 39
Participants | 1 | 0
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.30, Chi-squared

34. Secondary Outcome: Documented Myositis (PP)
Description: as for outcome 33
Time Frame: 54 Months Post-Randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 33 | 34
Participants | 1 | 0
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.31, Chi-squared

35. Secondary Outcome: Initiating Use of Disease-Modifying Antirheumatic Drugs (DMARDs) by Month 54 (ITT)
Description: Initiation of disease-modifying antirheumatic drugs (DMARDs). Participants were not expected to receive additional disease-modifying therapy for systemic sclerosis (SSc) in the absence of disease progression. In general, this includes the administration of any therapy clearly given for the purpose of treating the underlying SSc. It does not include concomitant treatments permitted in the protocol, such as use of methotrexate (15 g or less), anti-malarials, or minocycline for arthritis only. Systemic corticosteroids given at > 10 mg/day (prednisone or prednisone equivalent), without clearly defined non-SSc indications, and methotrexate given for non-arthritis indications are examples of qualifying DMARDs.
Time Frame: 54 Months Post-Randomization
Population: Intention to treat (ITT). The ITT population includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 36 | 39
Participants | 3 | 15
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.002, Chi-squared

36. Secondary Outcome: Initiating Use of Disease-Modifying Antirheumatic Drugs by Month 54 (DMARDs) (PP)
Description: as for outcome 35
Time Frame: 54 Months Post-Randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 33 | 34
Participants | 3 | 15
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.001, Chi-squared

37. Secondary Outcome: Regimen-Related Toxicities
Description: Regimen-related toxicities are defined as Grade 3 or higher adverse events reported by site physicians as possibly, probably, or definitely related to study therapy.
Time Frame: Randomization through end of study follow-up (up to Month 72 post-randomization)
Population: Safety population. The safety population includes all participants for whom study treatment was initiated. For the mHSCT arm, treatment was initiated with the first dose of granulocyte colony stimulating factor for mobilization, and for the cyclophosphamide arm, treatment was initiated with the first dose of IV cyclophosphamide.
Measure: Number; unit: Events
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 34 | 37
Events
  Possibly Related | 106 | 23
  Probably Related | 98 | 13
  Definitely Related | 90 | 5
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p < 0.001, Regression, Linear; P-value comes from a Poisson regression comparing the person-year adjusted event rates between the two treatment groups
Statistical Analysis 2: Comparison: mHSCT; Test type: Superiority; Person-Time (Years) = 174.4 — The Person-Time (P-T) rates (events/P-T) are as follows: Possibly related = 0.61, Probably related = 0.57, Definitely related = 0.52
Statistical Analysis 3: Comparison: Cyclophosphamide; Test type: Superiority; Person-Time (Years) = 141.3 — The Person-Time (P-T) rates (events/P-T) are as follows: Possibly related = 0.17, Probably related = 0.09, Definitely related = 0.04

38. Secondary Outcome: Number of Subjects With Regimen-Related Toxicities
Description: as for outcome 37
Time Frame: Randomization through end of study follow-up (up to Month 72 post-randomization).
Population: as for outcome 37
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 34 | 37
Participants
  Possibly Related | 33 | 10
  Probably Related | 27 | 10
  Definitely Related | 26 | 3

39. Secondary Outcome: Infectious Complications
Description: Infectious complications include any events that code to the Medical Dictionary for Regulatory Activities (MedDRA) system organ class of "Infections and infestations" or events that a site has classified as an infectious event. These can include bacteremia, septicemia, fungemia, fever associated with infection, infectious pneumonia, idiopathic pneumonia syndrome, clinical infection (i.e. infection diagnosed with clinical features without identification of an organism) and other local/organ site-specific infections.
Time Frame: Randomization through end of study follow-up (up to Month 72 post-randomization).
Population: as for outcome 37
Measure: Number; unit: Events
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 34 | 37
Events | 131 | 112
Statistical Analysis 1: Comparison: mHSCT vs Cyclophosphamide; Test type: Superiority; p = 0.7, Regression, Linear; P-value comes from a Poisson regression comparing the person-year adjusted event rates between the two treatment groups
Statistical Analysis 2: Comparison: mHSCT; Test type: Superiority; Person-Time (Years) = 174.4 — The Person-Time (P-T) rate (events/P-T) is 0.76
Statistical Analysis 3: Comparison: Cyclophosphamide; Test type: Superiority; Person-Time (Years) = 141.3 — The Person-Time (P-T) rate (events/P-T) is 0.80

40. Secondary Outcome: Number of Subjects With Infectious Complications
Description: as for outcome 39
Time Frame: Randomization through end of study follow-up (up to Month 72 post-randomization).
Population: as for outcome 37
Measure: Count of Participants; unit: Participants
Arm/Group | mHSCT | Cyclophosphamide
Number analyzed (Participants) | 34 | 37
Participants | 33 | 31

41. Secondary Outcome: Time to Absolute Neutrophil Count Engraftment
Description: Time to absolute neutrophil count (ANC) engraftment is defined as the number of days post-transplant until required levels of ANC are attained (for the mHSCT arm only). If engraftment did not occur within 28 days post-transplant, then the variable was set to 28 days. ANC engraftment required an ANC of > 500 cells/microliter, maintained for 3 consecutive days.
Time Frame: 28 days post-transplant
Population: Per-protocol (PP) - mHSCT arm only. The PP population is defined as those participants who completed the assigned treatment protocol: undergoing autologous CD34-selected hematopoietic progenitor cell transplantation in the mHSCT arm.
Measure: Median (Full Range); unit: Days
Arm/Group | mHSCT
Number analyzed (Participants) | 34
Days | 10 [8 to 12]

ADVERSE EVENTS:
Time Frame: From randomization until study completion, an average of 72 months, or until 30 days after a participant withdrew early from the study. All-cause mortality was additionally identified through site contact or public records after participant withdrawal.
Description: AEs were collected in the safety population (all participants for whom study treatment was initiated, defined as: mHSCT arm, first dose of granulocyte colony stimulating factor for mobilization; cyclophosphamide arm, first dose of IV cyclophosphamide). In the mHSCT arm, Grade 4 cytopenias reported that occur between conditioning and Day 28 after infusion of the IP are not reported as SAEs. All-cause mortality is reported in the ITT population (all randomized participants).
Arm/Group | mHSCT | Cyclophosphamide
All-Cause Mortality (participants affected / at risk) | 7/36 | 14/39
Serious Adverse Events (participants affected / at risk) | 25/34 | 19/37
Other Adverse Events (participants affected / at risk) | 33/34 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mHSCT (N=34) | Cyclophosphamide (N=37)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 4 (6) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 3 (4)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal hypomotility (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumatosis cystoides intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (4) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Heparin-induced thrombocytopenia (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (2)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Meningitis enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (6) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (4)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pulmonary function test decreased (Investigations) | 1 (1) | 4 (5)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dystonia (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Scleroderma renal crisis (Renal and urinary disorders) | 1 (1) | 3 (5)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Capillary leak syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mHSCT (N=34) | Cyclophosphamide (N=37)
Anaemia (Blood and lymphatic system disorders) | 19 (41) | 16 (23)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 26 (42) | 6 (15)
Lymphopenia (Blood and lymphatic system disorders) | 31 (73) | 25 (53)
Neutropenia (Blood and lymphatic system disorders) | 26 (34) | 4 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 29 (39) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 5 (6) | 2 (2)
Conjunctivitis (Eye disorders) | 3 (3) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (5)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 8 (16)
Diarrhoea (Gastrointestinal disorders) | 4 (7) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 6 (6) | 5 (5)
Gastritis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (6) | 5 (5)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 2 (3)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 6 (23)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 1 (2) | 2 (3)
Fatigue (General disorders) | 6 (8) | 5 (8)
Mucosal inflammation (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 5 (5) | 1 (1)
Bacteraemia (Infections and infestations) | 3 (3) | 0 (0)
Body tinea (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 2 (2)
Bronchitis acute (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 4 (4) | 2 (2)
Cystitis (Infections and infestations) | 2 (2) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 4 (4) | 0 (0)
Herpes zoster (Infections and infestations) | 11 (12) | 1 (1)
Infected skin ulcer (Infections and infestations) | 2 (4) | 4 (10)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 5 (12) | 2 (5)
Paronychia (Infections and infestations) | 2 (2) | 1 (2)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 3 (4) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 9 (14) | 8 (19)
Urinary tract infection (Infections and infestations) | 1 (2) | 11 (20)
Alanine aminotransferase increased (Investigations) | 9 (10) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 3 (3)
Ejection fraction decreased (Investigations) | 3 (3) | 1 (1)
Forced expiratory volume decreased (Investigations) | 11 (13) | 5 (5)
Pulmonary function test decreased (Investigations) | 23 (30) | 12 (16)
Vital capacity decreased (Investigations) | 6 (6) | 6 (6)
Weight decreased (Investigations) | 2 (2) | 6 (6)
Weight increased (Investigations) | 6 (6) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (6) | 2 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (9)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 (3) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 4 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (5)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (3)
Headache (Nervous system disorders) | 4 (6) | 5 (7)
Hypoaesthesia (Nervous system disorders) | 2 (3) | 3 (3)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (4) | 2 (2)
Depression (Psychiatric disorders) | 9 (11) | 8 (11)
Insomnia (Psychiatric disorders) | 5 (6) | 5 (6)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (4)
Proteinuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Vulvovaginal dryness (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (13) | 4 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 9 (9) | 2 (4)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 7 (14) | 10 (24)
Hot flush (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 2 (3) | 2 (2)
Hypotension (Vascular disorders) | 3 (6) | 2 (2)
Raynaud's phenomenon (Vascular disorders) | 4 (4) | 0 (0)

LIMITATIONS AND CAVEATS:
Results are applicable for SSc with severe internal organ disease and may not be generalizable to all those with dcSSc. The hierarchical components of the GRCS are specific to this SSc population and may not be generalizable to other SSc populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No